CLINICAL TRIAL: NCT01329172
Title: Impact of Polyunsaturated Fatty Acids n-3 on Nasal Mucins Expression in Cystic Fibrosis Patients
Brief Title: Nasal Mucin Oral Supplementation Treatment Respiratory Inflammation Using PUFA in Cystic Fibrosis (CF) Patients
Acronym: NOSTRIL
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2008_47/0928; 2009-014869-43 (EudraCT Number)
Record Dates: First submitted 2010-05-21; First posted 2011-04-05 (Estimated); Last update posted 2017-12-22 (Actual); Status verified 2017-12

CONDITIONS: Cystic Fibrosis; Dietary Modification
Keywords: PUFA; Cystic Fibrosis; Nasal brushing; Mucins; Mucin production
MeSH Terms: conditions — Cystic Fibrosis | interventions — Fatty Acids, Omega-3; Docosahexaenoic Acids

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- polyunsaturated fatty acids n-3 (Experimental): polyunsaturated fatty acids n-3 (PUFA n-3)
  Interventions: Other: polyunsaturated fatty acids n-3
- placebo (Placebo Comparator): sun flower oil
  Interventions: Other: placebo

INTERVENTIONS:
Other: polyunsaturated fatty acids n-3 — polyunsaturated fatty acids n-3 1 gram per day during two months
  Other Names: PUFA n-3
  Arms: polyunsaturated fatty acids n-3
Other: placebo — sun flower oil with Poly Unsaturated Fatty Acid 1g/day
  Other Names: PUFA
  Arms: placebo

SUMMARY:
Background :

Cystic fibrosis (CF) patients are prone to recurrent pulmonary infection have different secreted mucin pattern from healthy subjects. Long chain polyunsaturated fatty acids have been shown to influence survival and MUC5B expression in mice model of chronic pulmonary infection.

Method :

To study the impact of LCPUFA n-3 on MUC5B expression (mRNA level by RT-PCR) collected in airway epithelial cells obtained by nasal brushing. The secondary aim is to assess : MUC1, MUC2, MUC4, MUC5AC, MUC7 expression (mRNA level) in airway epithelial cells obtained by nasal brushing; Lund-Kennedy score; TNK-alpha, IL-6, IL-8 in blood plasma. This study is a double parallel, controlled double blind, randomized clinical trial : LCPUFA n-3 (1 g/day) vs placebo for 6 weeks. 30 subjects will be included in this study. Primary and secondary study end point will be assessed two times: before randomization and after 60 days of treatment.

Statistical analysis :

Treatment group and placebo will be compared using U-Mann-Whitney, intention to treat and per protocol.

DETAILED DESCRIPTION:
Primary Outcome Measure : Mucin MUC5B (mRNA level) in native airway epithelial cells obtained by nasal brushing

Secondary Outcome Measures : Mucin MUC1, MUC2, MUC4, MUC5AC, MUC7 (mRNA level) in native airway epithelial cells obtained by nasal brushing.

Lund-Kennedy score TNF-alpha, IL-6, IL-8 in plasma

ELIGIBILITY:
Inclusion Criteria :

* Cystic fibrosis patient
* Aged 18 to 30 year
* No modification of long term therapy (Corticoids, antibiotics, pancreatic extract, antiacid) before 4 weeks before randomization

Exclusion Criteria:

* Awaiting transplantation
* Patients on anticoagulants
* Contraindication to supplementation with polyunsaturated fatty acids
* Taking antibiotics in progress ( less than 15 days)
* Taking anti- inflammatory ongoing (more than one week per month , steroids , or nonsteroidal )

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2010-09-20 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Expression of Mucin "MUC5B" by measurement of messenger Ribo Nucleic Acid (mRNA) level in native airway epithelial cells obtained by nasal brushing | baseline and 2 months

SECONDARY OUTCOMES:
Mucin MUC1, MUC2, MUC4, MUC5AC, MUC7 (mRNA level) in native airway epithelial cells obtained by nasal brushing. Lund-Kennedy score TNF-alpha, IL-6, IL-8 in plasma | baseline and two months

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric GOTTRAND, MD, PhD, Study Chair — CHRU de Lille et Université Lille 2
Locations (3):
- France (3):
  - Dunkerque Hospital, Dunkirk
  - Lens Hospital, Lens
  - Clinical Investigation center, Lille

IPD SHARING:
Plan to Share IPD: No